CLINICAL TRIAL: NCT05405517
Title: Translation and Cross Cultural Validation on Modified Fatigue Impact Scale in Urdu Language
Brief Title: Translation of Modified Fatigue Impact Scale in Urdu Language
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: Fariha Zulfiqar
Record Dates: First submitted 2022-04-28; First posted 2022-06-06 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Traumatic Brain Injury
Keywords: Fatigue, TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cross cultural analytical study to translate Modified fatigue impact scale MFIS) in Urdu language. Along with the translated version by evaluating its validity and reliability among the patients of traumatic brain injury. No such study has been previously conducted in Pakistan which translate this scale in Urdu and follows the proper cross- culture adaptation.Condition or disease: Traumatic brain injury. Convenient sampling technique would be used.

DETAILED DESCRIPTION:
The MFIS is a modified version of 40-item Fatigue Impact Scale (FIS). The MFIS impact scale consist of 3 subdivisions containing 9 physical items , 10 cognitive items and 2 psychosocial. The maximum score is 84 which is obtained by the sum of all the questions The higher score means high impact on quality of life. This version should be answered by the patients with traumatic brain injury. It is the patient's self- report. As the MFIS is well- developed measurement scale, it is meaningful to translate and validate this scale in Urdu Version. It is useful the study the effect of fatigue in the patients with TBI by using same measurement items so that a more direct comparison can be made. Therefore, the aim of the study is to translate and validate the Modified Fatigue Impact scale in Urdu language The translation and cultural adaptation process would start after obtaining approval from the developer of the original MFIS. This would be done according to WHO guidelines. Translation will be done by symmetrical category. The purpose will be to gain uniformity in the translation of tool in both the Target language and source language. This will involve 5 steps. (Forward translation, synthesis 2, Backward translation, synthesis 2 and pilot testing). Phase 2 would be done according to the guidelines of COSMIN in which psychometric properties will be measured.(reliability, internal consistency, construct validity and factor analysis.)

ELIGIBILITY:
Inclusion Criteria

* Age 18-65 years
* Both Male and Female
* Patient Able to read Urdu Language
* Any period of loss of consciousness after 1 hour of injury
* Patients who can actively participate in community
* For comprehension patients with the MMSE score > 25 will be included

Exclusion Criteria:

* Patients able to perform 5 meter walk test
* Patients having score >6 in FIM scale
* For alcohol abuse patients with the score < 8 in AUDIT scale
* Any other neurological disease including Alzheimer, Parkinson's disease and Schizophrenia

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Traumatic Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Modified Fatigue impact scale | 8 months
  The modified fatigue impact scale consists of 21 questions. The version of MFIS questionnaire is divided into 3 subdivision containing 9 physical items , 10 cognitive items and 2 psychosocial. All the items are rated from 0-4 .
  The sum of all the questions are calculated where 84 is the highest score. Highest the score means higher the impact of fatigue in daily living.

SECONDARY OUTCOMES:
Reliability of translated versions of MFIS | 8 months
  To determine the reliability of cross-culturally adapted and translated MFIS in the patients with TBI .Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two intervals between different visits of the patient. Intra class correlation coefficient(ICC) will be determine for test retest reliability.
Validity of translated versions of MFIS | 8 months
  To determine the validity of cross-culturally adapted and translated MFIS in the patients with TBI. Validity is how accurate the results are. Thus this will be measured through various parameters to validate the translated versions as appropriate and applicable. Pearson correlation coefficient was used to find convergent validity. CVI will detremine to find Content Validity for Urdu translated tool.
  validity

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Mukhtar, MS, Principal Investigator — Riphah International University
Locations (1):
- Tehreem Mukhtar, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schiehser DM, Delano-Wood L, Jak AJ, Matthews SC, Simmons AN, Jacobson MW, Filoteo JV, Bondi MW, Orff HJ, Liu L. Validation of the Modified Fatigue Impact Scale in mild to moderate traumatic brain injury. J Head Trauma Rehabil. 2015 Mar-Apr;30(2):116-21. doi: 10.1097/HTR.0000000000000019. PMID 24413076
- [Background] Ziino C, Ponsford J. Measurement and prediction of subjective fatigue following traumatic brain injury. J Int Neuropsychol Soc. 2005 Jul;11(4):416-25. doi: 10.1017/s1355617705050472. PMID 16209422
- [Background] Khalil H, Al-Shorman A, Alghwiri AA, Abdo N, El-Salem K, Shalabi S, Aburub A. Cross cultural adaptation and psychometric evaluation of an Arabic version of the modified fatigue impact scale in people with multiple sclerosis. Mult Scler Relat Disord. 2020 Apr;39:101878. doi: 10.1016/j.msard.2019.101878. Epub 2019 Nov 29. PMID 31841967
- [Background] Hebert JR, Forster JE, Stearns-Yoder KA, Penzenik ME, Brenner LA. Persistent Symptoms and Objectively Measured Balance Performance Among OEF/OIF Veterans With Remote Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2018 Nov/Dec;33(6):403-411. doi: 10.1097/HTR.0000000000000385. PMID 29385020